CLINICAL TRIAL: NCT03794492
Title: Impact of Lymphocyte Anti-metabolite Immunosuppressions on Donor-Specific Anti-HLA Antibody and Kidney Graft Outcome: Open-label, Multi-center, Single Arm, Phase 4 Trial (DoSAKOM)
Brief Title: Impact of Lymphocyte Anti-metabolite Immunosuppressions on Donor-Specific Anti-HLA Antibody and Kidney Graft Outcome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 223KT17017
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-05

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Mycophenolic Acid; Tablets; Capsules; Tacrolimus; Methylprednisolone; Prednisolone; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mycophenolate mofetil (Experimental): One arm: Mycophenolate mofetil 500mg Tab. or 250mg Cap.
  Interventions: Drug: Mycophenolate mofetil 500mg Tab. or 250mg Cap.; Drug: Tacrolimus; Drug: Methylprednisolone/prednisolone; Drug: Basiliximab

INTERVENTIONS:
Drug: Mycophenolate mofetil 500mg Tab. or 250mg Cap. — - Orally, up to 1g BID(total 2g daily)
  Other Names: Myrept® Cap./Tab.
Drug: Tacrolimus — - Orally, check the blood ceocentration of tacrolimus at each visit and adjust the dose to acheive the blood concentration maintaining at 3-8ng/ml
Drug: Methylprednisolone/prednisolone — - Methyprednisolone 500mg / Prednisolone 5mg
Drug: Basiliximab — - IV, 20mg(before Kidney transplat) / 20mg(Day 4 of kidney transplant)

SUMMARY:
Efficacy and Safety of My-Rept® (Mycophenolate Mofetil 500mg/Tab. or 250mg/Cap.) in Combination with Tacrolimus, Methylprednisolone, Simulect in Kidney Transplant Patients

DETAILED DESCRIPTION:
This study is a multi-center, non-comparative and phase IV clinical trial that evaluates incidence of Donor-Specific Antibody for 36 months after kidney transplantation when administered with Tacrolimus, Mycophenolate mofetil, and corticosteroid

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old(male or female)
2. Patients who are planning to receive a kidney from a deceased or a living unrelated/related donor
3. Agreement with written informed consent

Exclusion Criteria:

1. Donor's HLA antigen matches recipient or the Degree of Mis-Match is 0
2. Patients with high sensitization who need desensitization therapy
3. Multi organ recipients or previous transplant with any organs
4. Diagnosed with cancer within five years
5. Patient who receive kidney from ABO incompatibility donor or Lymphocyte cross-match positive donor
6. Patients who have positive HIV, HBsAg or Anti-HCV test result
7. At screening

   * Under treatment for active liver disease, or Over 3times upper than normal range of liver function test (T-bilirubin, AST, ALT)
   * WBC<2,500/mm3, PLT <50,000/mm3, ANC<1,500/mm3
8. Pregnant or lactating women
9. In investigator's judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
DSA(Donor-specific Anti-HLA Antibody) | 36 months
  Incidence of DSA(Donor-specific Anti-HLA Antibody) up to 36months after Kidney transplantation

SECONDARY OUTCOMES:
Incidence of composite efficacy failure | 12, 24, 36months
  The frequency and percentage of composite efficacy failure (Treated-BPAMR & ACR, graft loss, death and follow-up loss)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Kwan Oh, Ph.D, Study Chair — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwan, South Korea

IPD SHARING:
Plan to Share IPD: No